CLINICAL TRIAL: NCT02459223
Title: Open Label Prospective Parallel Group Active Comparator Interventional Study to Determine the Efficacy of the Therapeutic Nutritional Intervention in SAM Category Malnourished Children of Satpuda Region.
Brief Title: Study of Blood Parameters of the Malnourished Children: Before and After Giving Nutritional Biscuit's Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharashtra University of Health Sciences (Other)
Responsible Party: Principal Investigator, Sangeeta Pingale, Open label prospective parallel group active comparator interventional study to determine the efficacy of the therapeutic nutritional intervention in SAM category malnourished children of satpuda region., Maharashtra University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NBT
Record Dates: First submitted 2015-05-19; First posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Undernutrition
Keywords: Nutritional intervention; iron deficiency anemia
MeSH Terms: conditions — Malnutrition; Anemia, Iron-Deficiency | interventions — Spices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Group (Active Comparator): Treated with nutritional biscuits and khichadi. Nutritional biscuits providing 2.5 to 3 gm Protein and 90-100kcal/kg body Weight/day, as well as local food Khichadi (Rice and hulled split green gram cooked together with spices) for the three months period.
  Interventions: Dietary Supplement: Nutritional biscuits and khichadi
- Control Group (Active Comparator): Treated with only local food Khichadi (Rice and hulled split green gram cooked together with spices) for the three months period.
  Interventions: Dietary Supplement: Khichadi

INTERVENTIONS:
Dietary Supplement: Nutritional biscuits and khichadi — Nutritional biscuits and Khichadi.
  Other Names: Khichadi means Rice cooked with lentiles and spices.
  Arms: Test Group
Dietary Supplement: Khichadi — Khichadi.
  Other Names: Khichadi means Rice cooked with lentiles and spices.
  Arms: Control Group

SUMMARY:
Present study was designed to evaluate the efficacy of the nutritional intervention, in the SAM (Severe Acute malnutrition)children by monitoring various Anthropometric,Biochemical ,Hormonal and Enzymatic parameters before and after the nutritional intervention treatment.This study was also intended to study possible functional role of gene HRI (heme regulated inhibitor) as a molecular marker for the early detection of iron deficiency anemia in malnourished children similarly present study has also tried to find anthropometric marker and different correlations among study parameters.

DETAILED DESCRIPTION:
In India, child malnutrition is responsible for 22% of the country's burden of disease. Development of local therapeutic nutritional intervention is highly recommended by WHO. Present study was designed to evaluate the efficacy of the nutritional intervention, as well as to study HRI (heme regulated inhibitor) gene expression, to suggest it as a molecular marker for the early detection of iron deficiency anemia in malnourished children also to find anthropometric marker and different correlations of study parameters.

105 test and 100 control SAM (Severe Acute malnutrition) children without infection, of 1 to 5 years of age and either sex were enrolled. Test group was given treatment of nutritional intervention therapy (NIT), providing 2.5 to 3gm Protein and 90-100kcal/kg body Weight/day, for the three months period. Their Anthropometric, Enzymatic, Biochemical and Hormonal parameters were measured before and after the NIT. Correlation of serum triglyceride with weight for height% , as well as correlation of HRI with Mean corpuscular hemoglobin,(MCH) was studied. Similarly status of Hairs, Skin, oedema, WHO z- score,and BMR was also studied before and after the NIT.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from age group of 1 to 5 years of either sex belonging to SAM (Severe Acute Malnutrition) category and provided Therapeutic Nutritional Biscuit's treatment.
* Subjects from age group of 1 to 5 years of either sex belonging to SAM and not taking nutritional Biscuit's treatment, included as a control for comparative study.

Exclusion Criteria:

* Children above 5 years of either sex.
* SAM children with various infections.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Measurement of Anthropometric Parameters as a measure of improvement in malnutrition. | 3 months
  All the enrolled test group malnourished children have put on weight at a rate of 5 g/kg/day and their WHO z-score for weight and Height were improved from -3 to -1 Or Normal, as well as MUAC improved to normal and edema was absent.
Measurement of biochemical Parameters as a measure of improvement in malnutrition. | 3 months.
  The level of all blood parameters were noted to be improved from abnormal to normal level in the all enrolled test group malnourished children.
Measurement of expression of gene HRI (Heme Regulatory Inhibitor) as a measure of improvement in iron storage and malnutrion. | 3 months
  The expression of Gene HRI was noted to be down regulated in the all enrolled test group malnourished children.

SECONDARY OUTCOMES:
Correlations among Anthropometric,Blood and Genetic parameters as a measure of strong or weak relationship. | 3 months
  There were improvements noted in the Anthropometric and Blood parameters,Gene HRI was also noted to be down-regulated
ANOVA test and Regression as a measures of statistical marker. | 3 months
  Two markers were proposed.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Pingale, Ph.D.appear, Principal Investigator — Maharashtra University of Health Sciences,nashik,Maharashtra,India
Locations (1):
- Sangeeta Pingale, Nashik, Maharashtra, India